CLINICAL TRIAL: NCT07048444
Title: Data Collection for a Surface Caries Detection Software
Brief Title: Surface Caries Feature Study
Status: Not yet recruiting | Type: Observational
Sponsor: 3Shape A/S (Industry)
Collaborators: New York University (Other)
Responsible Party: Sponsor
Other Study IDs: CIS-004
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Caries Active; Caries Root; Caries,Dental; Caries; Initial; Caries Assessment
MeSH Terms: conditions — Root Caries; Dental Caries | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Caries active patients: Patients with a history of caries
  Interventions: Other: N/A as observational study

INTERVENTIONS:
Other: N/A as observational study — N/A as observational study design

SUMMARY:
Dental caries (dental cavity) is very common and can impact oral health and oral health-related quality of life. Dental caries is when the tooth surfaces break down, and if left untreated, can cause tooth pain. In routine clinical practice, dental professionals typically assess caries lesions by looking at patients' teeth, touching the areas of interest with a dental probe, and running a probe over the teeth to check the buildup of bacteria.

Dentists often use x-rays to help find cavities, and they can also take pictures of the teeth to show what the problem looks like.

New tools called intraoral scanners are becoming more useful for finding cavities. These scanners do not use radiation and do not hurt. Some computer programs that use artificial intelligence (AI) can also help dentists find cavities. AI can study the spots on patients' teeth and help make better, faster decisions. The purpose of this study is to collect data that will be used to develop and test an AI software that can help dentists in the detection of caries.

DETAILED DESCRIPTION:
This is a single-arm, cross-sectional, open single-site clinical investigation using TRIOS 5 and TRIOS 6 intraoral scanners.

After enrolment, the participant will first undergo an intraoral scan. Next, the participant's teeth will be cleaned to remove plaque and debris, ensuring optimal conditions for the caries examination. Dental bitewing radiographs will be taken to assess any potential caries not visible on the scan. A second intraoral scan will be performed on the cleaned teeth. The examiner will then conduct an examination using standardized diagnostic criteria to assess the presence of caries, and will take intraoral photos of the caries lesions.

The AI-based software will provide a digital assessment of caries for comparison with the clinical evaluation. This comparison will be conducted separately from the clinical data collection. The comparison of the AI output to the clinical data will be performed internally at 3Shape headquarters of Holmens Kanal 7, 1060, Copenhagen, Denmark. This test has no impact on the patients in this study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Male or female, aged 18 years or above
* Patients looking for dental treatment
* Good general health (i.e. absence of any condition that the Principal Investigator evaluates as a risk either to the subject or to the data quality)
* Able (in the Investigator's opinion) and willing to comply with all study requirements.
* Minimum of 15 natural teeth without crowns
* At least one cavitated caries lesion

Exclusion Criteria:

* Patients with orthodontic appliances and permanent retainers
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study)
* Patients who are not able or willing to sign the Informed Consent
* Patients who are currently pregnant. A urine pregnancy test will be administered during the study visit for woman who could be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants, representing a cross-section of the general population of those persons that seek dental treatment, will be recruited according to an age span from 18 years and above
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2025-07-22 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy for surface caries detection software (SCDS) in surface caries detection on visible tooth surfaces compared to clinical visual tactile examination using the International Caries Detection and Assessment System (ICDAS) | Baseline
  Sensitivity of ≥0.68 and specificity of ≥0.83 for SCDS diagnostic accuracy in surface caries detection on visible tooth surfaces compared to clinical visual tactile examination using the ICDAS